CLINICAL TRIAL: NCT00892242
Title: Perioperative Treatment With Zoledronic Acid in Patients With Resectable Pancreas Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Principal Investigator decided to close the study early.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0589 / 201109094
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Adenocarcinoma
Keywords: Neoadjuvant zoledronic acid in resectable pancreas cancer
MeSH Terms: conditions — Adenocarcinoma | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neoadjuvant Zoledronic Acid (Experimental): Zoledronic acid 4 mg IV prior to pancreatic resection (approximately 2 weeks prior to resection)
  Pancreatic resection
  Zoledronic acid 4 mg IV monthly for two additional doses
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid
  Other Names: Zometa

SUMMARY:
The overall purpose of this research is to evaluate the safety and side effects of zoledronic acid (also known as Zometa) in patients before they have surgery to remove the cancer.

DETAILED DESCRIPTION:
Cancer of the pancreas carries an ominous prognosis. The five-year overall survival rate of this malignancy is less than 5%. Chemotherapy with gemcitabine carries a response rate of approximately 25%. Resection offers the only potential for cure; however, even with resection, the great majority of patients will die with metastatic disease. Substantial improvements are needed in the treatment of this malignancy.

Patients with this disease process have clearly developed a tolerance to their pancreatic tumor. This is evidenced by an increased number and activity immunosuppressive cells including MDSC and Treg in patients with pancreas cancer. An intervention that inhibits this population of MDSC and Treg may be highly useful in the treatment of this disease process.

A novel treatment of pancreas cancer, in this setting, would be to deplete circulating and tumor-associated immunosuppressive cells prior to resection. This would facilitate the host to mount a greater immune response against the tumor. The eventual goal would be to combine neoadjuvant zoledronic acid with gemcitabine, another agent which synergizes with zoledronic acid to target MDSC. When combined with current adjuvant chemoradiation, the use of zoledronic acid in the neoadjuvant and adjuvant setting, it is hoped that the patient could mount a greater immune response leading to increased overall survival through the prevention of local disease and distant metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a newly diagnosed, histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma. The histological slides or blocks must be available for review.
* Patient must have resectable disease and be a candidate for surgical treatment.
* Recent CT scan demonstrating pancreatic tumor, no evidence of distant disease, and no contraindication to resection.
* Patients must be ≥ 18 years old.
* Performance Status: Karnofsky Performance Status (KPS) ≥ 70
* Life Expectancy > 12 weeks.
* No previous history of chemotherapy for pancreas cancer prior to the start of protocol treatment.
* Patients must have recovered from uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
* Patients must have adequate bone marrow function defined as an absolute neutrophil count >1,500/mm3, platelet count >100,000/mm3 and hemoglobin >10 g/dl.
* Patients must have normal renal function defined as serum creatinine ≤ 1.3 mg/dl or creatinine clearance ≥ 90 ml/min/1.73 m2 with a serum creatinine > 1.3 mg/dl.
* Patients must have adequate hepatic function with total bilirubin < 5.0 mg/dl and AST ≤ 3x the institutional normal value.
* Patient must have no prior or current active autoimmune disease requiring management with immunosuppression. This includes inflammatory bowel disease, systemic vasculitis, scleroderma, psoriasis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjogren's syndrome, sarcoidosis or other rheumatologic disease. Asthma and chronic obstructive pulmonary disease that does not require daily systemic corticosteroids is acceptable.
* The patient with previous history of malignancy is eligible for this study only if the patient meets the following criteria for cancer survivor: (i) patient has undergone potentially curative therapy for all prior malignancies; (ii) the patient has been considered disease free for at least 5 years; (iii) adequately treated non-melanomatous skin cancer.
* For all sexually active patients, the use of adequate barrier contraception (hormonal or barrier method of birth control) will be required during therapy, prior to study entry and for the duration of study participation. Non-pregnant status will be determined in all women of childbearing potential.
* After being informed of the treatment involved, patients (or their legally authorized representative) must given written consent.

Exclusion Criteria:

* Patient is currently receiving other investigational agents.
* Pregnant and nursing women patients are not eligible.
* Patients known to be HIV positive are ineligible because of the potential inability to modulate immune responses (patient self-report).
* Patients treated with any bisphosphonate-based therapeutic for any indication, during the previous year.
* Patients with recent (within 6 weeks) or planned dental or jaw surgery dental or jaw surgery (e.g. extraction, implants).
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
* Patients with a history of aspirin sensitive asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-12; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and feasibility perioperative neoadjuvant zoledronic acid in patients with resectable pancreas cancer. | 1 year postoperatively
  Rate of grade 3 and 4 toxicities, especially nephrotoxicity, electrolyte imbalance and osteonecrosis of the jaw.
Evaluate whether treatment with perioperative zoledronic acid prolongs overall survival or disease free survival. | 2 years

SECONDARY OUTCOMES:
Determine the pharmacodynamics on selected immune cell subgroups in the peripheral blood and marrow by flow cytometric analysis. | Marrow (prior to first dose of zoledronic acid and week 10), peripheral blood (prior to first dose of zoledronic acid, week 10, and month 6)
Determine the pharmacodynamics of neoadjuvant zoledronic acid therapy on selected immune cell subgroups in the tumor microenvironment by flow cytometric analysis of pancreatic tumor samples. | Approximately week 2 (at time of surgery)
Determine the pharmacodynamics of neoadjuvant zoledronic acid therapy on the neoangiogenesis. | Prior to zoledronic acid treatment and then completion of zoledronic acid treatment (approximately 10 weeks)
  Surrogate markers of tumor-associated neoangiogenesis will be analyzed by ELISA. Serum levels of VEGF and MMP9 will be measured compared pre and post treatment.
Determine the pharmacodynamics and surrogate markers neoangiogenesis analyzed by ELISA. | Prior to zoledronic acid treatment and then completion of zoledronic acid treatment (approximately 10 weeks)
  Serum levels of VEGF and MMP9 will be measured compared pre and post treatment and the expression of VEGF and MMP9 in tumor samples will be analyzed.
Measure the presence and change of micrometastatic disease present in the bone marrow at the time of surgery versus baseline using immunohistochemistry. | Baseline and week 2 (time of surgery)
Evaluate the clinical response and time to disease progression. | 6 months postoperatively
Correlate the presence of micrometastatic disease with time to recurrence and outcome. | 6 months postoperatively
Measure the change in the amount of micrometastatic disease from baseline. | 6 months postoperatively
Determine the pharmacodynamics of neoadjuvant zoledronic acid therapy on selected immune cell subgroups in the hepatic metastatic niche by flow cytometric analysis of pancreatic tumor samples | Approximately 2 weeks (time of surgery)

CONTACTS AND LOCATIONS:
Overall Officials: David Linehan, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Moore MJ, Goldstein D, Hamm J, Figer A, Hecht JR, Gallinger S, Au HJ, Murawa P, Walde D, Wolff RA, Campos D, Lim R, Ding K, Clark G, Voskoglou-Nomikos T, Ptasynski M, Parulekar W; National Cancer Institute of Canada Clinical Trials Group. Erlotinib plus gemcitabine compared with gemcitabine alone in patients with advanced pancreatic cancer: a phase III trial of the National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 2007 May 20;25(15):1960-6. doi: 10.1200/JCO.2006.07.9525. Epub 2007 Apr 23. PMID 17452677
- [Background] Gabrilovich DI, Bronte V, Chen SH, Colombo MP, Ochoa A, Ostrand-Rosenberg S, Schreiber H. The terminology issue for myeloid-derived suppressor cells. Cancer Res. 2007 Jan 1;67(1):425; author reply 426. doi: 10.1158/0008-5472.CAN-06-3037. No abstract available. PMID 17210725
- [Background] Linehan DC, Tan MC, Strasberg SM, Drebin JA, Hawkins WG, Picus J, Myerson RJ, Malyapa RS, Hull M, Trinkaus K, Tan BR Jr. Adjuvant interferon-based chemoradiation followed by gemcitabine for resected pancreatic adenocarcinoma: a single-institution phase II study. Ann Surg. 2008 Aug;248(2):145-51. doi: 10.1097/SLA.0b013e318181e4e9. PMID 18650621
- [Background] Varadhachary GR, Wolff RA, Crane CH, Sun CC, Lee JE, Pisters PW, Vauthey JN, Abdalla E, Wang H, Staerkel GA, Lee JH, Ross WA, Tamm EP, Bhosale PR, Krishnan S, Das P, Ho L, Xiong H, Abbruzzese JL, Evans DB. Preoperative gemcitabine and cisplatin followed by gemcitabine-based chemoradiation for resectable adenocarcinoma of the pancreatic head. J Clin Oncol. 2008 Jul 20;26(21):3487-95. doi: 10.1200/JCO.2007.15.8642. PMID 18640929
- [Background] Almand B, Clark JI, Nikitina E, van Beynen J, English NR, Knight SC, Carbone DP, Gabrilovich DI. Increased production of immature myeloid cells in cancer patients: a mechanism of immunosuppression in cancer. J Immunol. 2001 Jan 1;166(1):678-89. doi: 10.4049/jimmunol.166.1.678. PMID 11123353
- [Background] Schmielau J, Finn OJ. Activated granulocytes and granulocyte-derived hydrogen peroxide are the underlying mechanism of suppression of t-cell function in advanced cancer patients. Cancer Res. 2001 Jun 15;61(12):4756-60. PMID 11406548
- [Background] Diaz-Montero CM, Salem ML, Nishimura MI, Garrett-Mayer E, Cole DJ, Montero AJ. Increased circulating myeloid-derived suppressor cells correlate with clinical cancer stage, metastatic tumor burden, and doxorubicin-cyclophosphamide chemotherapy. Cancer Immunol Immunother. 2009 Jan;58(1):49-59. doi: 10.1007/s00262-008-0523-4. Epub 2008 Apr 30. PMID 18446337
- [Background] Melani C, Sangaletti S, Barazzetta FM, Werb Z, Colombo MP. Amino-biphosphonate-mediated MMP-9 inhibition breaks the tumor-bone marrow axis responsible for myeloid-derived suppressor cell expansion and macrophage infiltration in tumor stroma. Cancer Res. 2007 Dec 1;67(23):11438-46. doi: 10.1158/0008-5472.CAN-07-1882. PMID 18056472
- [Background] Tassone P, Tagliaferri P, Viscomi C, Palmieri C, Caraglia M, D'Alessandro A, Galea E, Goel A, Abbruzzese A, Boland CR, Venuta S. Zoledronic acid induces antiproliferative and apoptotic effects in human pancreatic cancer cells in vitro. Br J Cancer. 2003 Jun 16;88(12):1971-8. doi: 10.1038/sj.bjc.6600986. PMID 12799645
- [Background] Marten A, Lilienfeld-Toal Mv, Buchler MW, Schmidt J. Zoledronic acid has direct antiproliferative and antimetastatic effect on pancreatic carcinoma cells and acts as an antigen for delta2 gamma/delta T cells. J Immunother. 2007 May-Jun;30(4):370-7. doi: 10.1097/CJI.0b013e31802bff16. PMID 17457212
- [Background] Giraudo E, Inoue M, Hanahan D. An amino-bisphosphonate targets MMP-9-expressing macrophages and angiogenesis to impair cervical carcinogenesis. J Clin Invest. 2004 Sep;114(5):623-33. doi: 10.1172/JCI22087. PMID 15343380
- [Background] Santini D, Vincenzi B, Galluzzo S, Battistoni F, Rocci L, Venditti O, Schiavon G, Angeletti S, Uzzalli F, Caraglia M, Dicuonzo G, Tonini G. Repeated intermittent low-dose therapy with zoledronic acid induces an early, sustained, and long-lasting decrease of peripheral vascular endothelial growth factor levels in cancer patients. Clin Cancer Res. 2007 Aug 1;13(15 Pt 1):4482-6. doi: 10.1158/1078-0432.CCR-07-0551. PMID 17671133
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu